CLINICAL TRIAL: NCT04777500
Title: Applying Transcutaneous Auricular Vagus Nerve Stimulation to Treat Fibromyalgia
Brief Title: taVNS Treatment for Fibromyalgia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jian Kong, Principle investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020P003800
Record Dates: First submitted 2021-02-17; First posted 2021-03-02 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Fibromyalgia
Keywords: taVNS; Pain; Neuromodulation; Fibromyalgia
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- taVNS Group1 (Experimental): This group will receive taVNS for 4 weeks.
  Interventions: Device: Auricular transcutaneous electrical nerve stimulation device
- taVNS Group 2 (Experimental): This group will receive taVNS for 4 weeks.
  Interventions: Device: Auricular transcutaneous electrical nerve stimulation device

INTERVENTIONS:
Device: Auricular transcutaneous electrical nerve stimulation device — We are investigating whether taVNS can relieve chronic pain symptoms associated with Fibromyalgia.

SUMMARY:
In this research study we want to learn more about if transcutaneous electrical nerve stimulation (TENS), a safe electrical stimulation tool, can relieve Fibromyalgia pain. A total of 60 subjects with Fibromyalgia will be enrolled in this study at Massachusetts General Hospital, Charlestown Navy Yard campus.

ELIGIBILITY:
Inclusion Criteria:

* Meet the American College of Rheumatology (ACR) 1990 classification criteria and the ACR 2010 diagnostic criteria for fibromyalgia as determined by clinicians.
* Willingness to complete a 4-week, twice-a-day treatments.
* At least a 10th grade English-reading level; English can be a second language provided that the patients understand all questions used in the assessment measures.

Exclusion Criteria:

* Diagnosed with medical conditions that are known to contribute to fibromyalgia symptomatology, such as thyroid disease, inflammatory arthritis, systemic lupus erythematosus, rheumatoid arthritis, myositis, vasculitis, or Sjogren's syndrome.
* History of cardiac, respiratory, or nervous system disease that, in the investigator's judgment, precludes participation in the study because of a heightened potential for adverse outcome. For example: asthma or claustrophobia.
* Personal history of medical or psychiatric illness as determined by investigator.
* Pregnant or lactating.
* Less than a 10th grade English-reading level; English can be a second language provided that the patients understand all questions used in the assessment measures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Revised Fibromyalgia Impact Questionnaire (FIQR) | Baseline, week 2 and week 4.
  A change in the FIQR would indicate that participants are experiencing pain relief.

SECONDARY OUTCOMES:
Patient Reported Outcomes Measurement Information System (PROMIS-29) | Baseline, week 2 and week 4.
Pain Catastrophizing Scale | Baseline, week 2 and week 4.
Beck Depression Inventory-II (BDI-II) | Baseline and week 4.
Brief Quantitative Sensory Testing (QST) | Baseline and week 4.
Heart rate variability | Baseline and week 4.
power of oscillations in the alpha, theta, and gamma frequencies (optional) | Baseline and week 4.
  6 minutes of resting state EEG (with eyes open) (Optional). We will calculate the power of oscillations in the alpha, theta, and gamma frequencies, which will be normalized by the mean power for the global spectrum.
Blood inflammation markers (optional) | Baseline and week 4
  We will examine inflammatory mediators such as interleukins (ILs including IL-1β, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, and IL-10), IFN-γ, and tumor necrosis factor (TNF) via multiplex immunoassays using Luminex, as well as highly sensitive C-reactive protein (hsCRP), programmed death 1 (PD-1), prostaglandin E2, and BDNF.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Kong, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No